CLINICAL TRIAL: NCT03220737
Title: A Phase 4 Study to Assess the Safety and Immunogenicity of VAXCHORA (Cholera Vaccine, Live, Oral) in Children 2 to <18 Years of Age
Brief Title: VAXCHORA Pediatric Study to Assess Safety and Immunogenicity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Collaborators: Emergent BioSolutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PXVX-VC-200-006
Record Dates: First submitted 2017-07-11; First posted 2017-07-18 (Actual); Results first posted 2020-11-19 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Cholera (Disorder)
MeSH Terms: conditions — Cholera | interventions — Vaxchora; Cholera Vaccines

STUDY DESIGN:
Intervention Model Description: This is a randomized, placebo-controlled, double-blind, single-crossover study with three age cohorts and two treatment groups within each cohort.
  The main study consists of a screening period of 30 days, a treatment period from Day 1 to Day 29, and a follow-up period through Day 181. Cohort 1 has an optional sub-study consisting of a long-term follow-up period through Day 730.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will be conducted as a double-blind study through 181, where neither the sponsor, the statistical team, study volunteer subjects, nor clinical site personnel (except for the unblinded administration staff) will know subjects' treatment assignment. Once each subject has reached their Day 181 visit they will be individually unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort 1 (active, 12-17 yrs) (Experimental): Subjects aged 12 - 17 were administered a 100 mL oral dose of Vaxchora vaccine on Day 1, and had study visits on Day 11, 29, 91 and 181. Cohort 1 subjects that continued in the long-term follow-up sub-study had visits on days 365, 547 and 730.
  Interventions: Biological: VAXCHORA (Cholera Vaccine, Live, Oral)
- Cohort 1 (placebo, 12 - 17 yrs) (Placebo Comparator): Subjects aged 12 - 17 were administered a 100 mL oral dose of 0.9% saline on Day 1, and had study visits on Day 11, 29, 91 and 181.
  Interventions: Other: Placebo
- Cohort 2 (active, 6 - 11 yrs) (Experimental): Subjects aged 6 - 11 were administered a 100 mL oral dose of Vaxchora vaccine on Day 1, and had study visits on Day 11, 29, 91 and 181.
  Interventions: Biological: VAXCHORA (Cholera Vaccine, Live, Oral)
- Cohort 2 (placebo, 6 - 11 yrs) (Placebo Comparator): Subjects aged 6 - 11 were administered a 100 mL oral dose of 0.9% saline on Day 1, and had study visits on Day 11, 29, 91 and 181.
  Interventions: Other: Placebo
- Cohort 3 (active, 2 - 5 yrs) (Experimental): Subjects aged 2 - 5 were administered a 50 mL oral dose of Vaxchora vaccine on Day 1, and had study visits on Day 11, 29, 91 and 181.
  Interventions: Biological: VAXCHORA (Cholera Vaccine, Live, Oral)
- Cohort 3 (placebo, 2 - 5 yrs) (Placebo Comparator): Subjects aged 2-5 were administered a 50 mL oral dose of 0.9% saline on Day 1, and had study visits on Day 11, 29, 91 and 181.
  Interventions: Other: Placebo
- Historical Control: Adult Bridging Population (Other): This arm consists of historical data from Vaxchora vaccine subjects from study PXVX-VC-200-004. The data was included in study PXVX-VC-200-006 as a comparator bridging population for the Day 11 seroconversion. NCT02094586 PubMed ID:29317118
  Interventions: Biological: VAXCHORA (Cholera Vaccine, Live, Oral)

INTERVENTIONS:
Biological: VAXCHORA (Cholera Vaccine, Live, Oral) — VAXCHORA (Cholera Vaccine, Live, Oral) is a live, attenuated bacterial vaccine suspension for oral administration containing the V. cholerae strain CVD 103-HgR.
  Arms: Cohort 1 (active, 12-17 yrs); Cohort 2 (active, 6 - 11 yrs); Cohort 3 (active, 2 - 5 yrs); Historical Control: Adult Bridging Population
Other: Placebo — Placebo control for this study is normal (0.9%) saline.
  Arms: Cohort 1 (placebo, 12 - 17 yrs); Cohort 2 (placebo, 6 - 11 yrs); Cohort 3 (placebo, 2 - 5 yrs)

SUMMARY:
VAXCHORA (Cholera Vaccine, Live, Oral) is a vaccine indicated for active immunization against disease caused by Vibrio cholerae serogroup O1. VAXCHORA is approved for use in adults 18 through 64 years of age travelling to cholera-affected areas. The primary goals of this Phase 4 study are to evaluate the safety and immunogenicity of a single dose of VAXCHORA (1 x 10e9 cfu/dose) in children ages 2 years to <18 years of age in developed countries.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind, single-crossover study with three age cohorts and two treatment groups within each cohort.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Between 2 and <18 years of age on Day 1
* In general good health
* Able and willing to provide informed assent for study participation
* Primary caregiver is able and willing to provide informed consent for study participation
* (for females of childbearing potential) Using an acceptable method of contraception through Day 29

Exclusion Criteria:

* Current acute gastrointestinal illness or loose stools within 3 days of Day 1 visit
* Current acute febrile illness
* History of cholera infection
* History of cholera vaccination
* History of severe allergic reaction (e.g. anaphylaxis) to any ingredient of VAXCHORA
* Congenital or acquired immunodeficiency
* Pregnancy (for females of childbearing potential)
* Any other condition that, in the opinion of the Investigator, creates an unacceptable risk to the subject
* Any other condition that, in the opinion of the Investigator, will interfere with the conduct of the study or the validity of the data
* Duration of >2 weeks of abnormal stool pattern, defined as <3 stools per week or >2 stools per day in the past 6 months
* Regular use of laxatives in the past 6 months
* History of enterotoxigenic E. coli infection
* Travel to cholera-endemic area in the previous 5 years
* Nursing/Breastfeeding
* Received or plans to receive the following from 14 days prior to the study vaccination through 11 days after vaccination: Any other licensed vaccines, antibiotics, or chloroquine
* Received or plans to receive any other investigational agent throughout the main study (Day 181)

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 550 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2020-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Andre de Lame, MD, Study Director — Emergent BioSolutions
Locations (10):
- United States (10):
  - Emory University, Atlanta, Georgia
  - Johnson County Clin-Trials, Inc., Lenexa, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Boston Medical Center, Boston, Massachusetts
  - The Center for Pharmaceutical Research, Kansas City, Missouri
  - Rochester Clinical Research, Inc., Rochester, New York
  - Aventiv Research Inc., Columbus, Ohio
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Clinical Research Associates, Inc., Nashville, Tennessee

REFERENCES:
- [Derived] McCarty JM, Gierman EC, Bedell L, Lock MD, Bennett S. Safety and Immunogenicity of Live Oral Cholera Vaccine CVD 103-HgR in Children and Adolescents Aged 6-17 Years. Am J Trop Med Hyg. 2020 Jan;102(1):48-57. doi: 10.4269/ajtmh.19-0241. PMID 31769402

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study included healthy volunteers (2 - 17 years) who were not previously immunized against cholera. A total of 574 subjects were screened, of which 24 were screen failures. A total of 550 subjects randomized, of which 471 received study treatment and 433 and 73 completed the main study for treatment and placebo, respectively. Recruitment July 2017-July 2018.
Pre-assignment Details: This study included healthy volunteers (2 - 17 years) who were not previously immunized against cholera. A total of 574 subjects were screened, of which 24 were screen failures. A total of 550 subjects randomized, of which 471 received study treatment and 506 and 62 completed the main and sub studies, respectively. Recruitment July 2017-July 2018.
  The historical control subjects are not included in the protocol enrollment number for PXVX-VC-200-006. They are solely a comparator population.
Period: Main Study (Day 1 - 181)
Arm/Group | Cohort 1 (Active, 12-17 Yrs) | Cohort 1 (Placebo, 12 - 17 Yrs) | Cohort 2 (Active, 6 - 11 Yrs) | Cohort 2 (Placebo, 6 - 11 Yrs) | Cohort 3 (Active, 2 - 5 Yrs) | Cohort 3 (Placebo, 2 - 5 Yrs) | Historical Control: Adult Bridging Population
Started | 163 | 26 | 158 | 27 | 150 | 26 | 2688
Completed | 157 | 24 | 146 | 24 | 130 | 25 | 2687
Not Completed | 6 | 2 | 12 | 3 | 20 | 1 | 1
Not completed — Withdrawal by Subject | 4 | 1 | 4 | 1 | 4 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 6 | 1 | 13 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 1 | 3 | 0 | 1
Not completed — Failed Exl 8 and randomized in error | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Placebo Crossover (Day 181-365)
Arm/Group | Cohort 1 (Active, 12-17 Yrs) | Cohort 1 (Placebo, 12 - 17 Yrs) | Cohort 2 (Active, 6 - 11 Yrs) | Cohort 2 (Placebo, 6 - 11 Yrs) | Cohort 3 (Active, 2 - 5 Yrs) | Cohort 3 (Placebo, 2 - 5 Yrs) | Historical Control: Adult Bridging Population
Started | 13 (Only placebo subjects who opted to receive Vaxchora were included in the crossover group.) | 0 (Placebo subjects from Main study opted to cross over to the active group to receive Vaxchora.) | 11 (Only placebo subjects who opted to receive Vaxchora were included in the crossover group.) | 0 (Placebo subjects from Main study opted to cross over to the active group to receive Vaxchora) | 7 (Only placebo subjects who opted to receive Vaxchora were included in the crossover group.) | 0 (Placebo subjects from Main study opted to cross over to the active group to receive Vaxchora) | 0
Completed | 13 | 0 | 11 | 0 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 2 | 0 | 0
Period: Long-term Follow-up (Day 365-730)
Arm/Group | Cohort 1 (Active, 12-17 Yrs) | Cohort 1 (Placebo, 12 - 17 Yrs) | Cohort 2 (Active, 6 - 11 Yrs) | Cohort 2 (Placebo, 6 - 11 Yrs) | Cohort 3 (Active, 2 - 5 Yrs) | Cohort 3 (Placebo, 2 - 5 Yrs) | Historical Control: Adult Bridging Population
Started | 73 (Cohort 1 subjects from the main study had to opt to be included in the Long-term follow-up study.) | 0 | 0 (Cohort 2 subjects were not eligible for the Long-term follow-up study.) | 0 | 0 (Cohort 3 subjects were not eligible for the Long-term follow-up study.) | 0 | 0
Completed | 62 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 11 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 9 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Subject did not want lab drawn | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Historical Control: Adult Bridging Population: This arm consists of historical data from Vaxchora vaccine subjects from study PXVX-VC-200-004. The data was included in study PXVX-VC-200-006 as a comparator bridging population for the Day 11 seroconversion. NCT02094586, PubMed ID: 29317118
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Active, 12-17 Yrs) | Cohort 1 (Placebo, 12 - 17 Yrs) | Cohort 2 (Active, 6 - 11 Yrs) | Cohort 2 (Placebo, 6 - 11 Yrs) | Cohort 3 (Active, 2 - 5 Yrs) | Cohort 3 (Placebo, 2 - 5 Yrs) | Historical Control: Adult Bridging Population | Total
Number analyzed (Participants) | 163 | 26 | 158 | 27 | 150 | 26 | 2688 | 3238
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 163 | 26 | 158 | 27 | 150 | 26 | 0 | 550
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 2688 | 2688
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.4 (1.7) | 14.3 (1.7) | 8.6 (1.8) | 8.7 (1.5) | 3.5 (1.1) | 3.6 (1.2) | 30.0 (7.8) | 9.0 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 12 | 81 | 10 | 69 | 17 | 1482 | 1746
  Male | 88 | 14 | 77 | 17 | 81 | 9 | 1206 | 1492
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1 | 1 | 0 | 11 | 14
  Asian | 1 | 0 | 4 | 0 | 0 | 0 | 56 | 61
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8
  Black or African American | 28 | 4 | 53 | 5 | 67 | 14 | 671 | 842
  White | 121 | 21 | 86 | 18 | 71 | 12 | 1855 | 2184
  More than one race | 13 | 0 | 15 | 3 | 11 | 0 | 50 | 92
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 37 | 37
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 163 | 26 | 158 | 27 | 150 | 26 | 2341 | 2891
  Australia | 0 | 0 | 0 | 0 | 0 | 0 | 347 | 347

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1 (12-17 Yrs) Primary Endpoint - Seroconversion of Serum Vibriocidal Antibody Against V. Cholerae
Description: The proportion of subjects achieving seroconversion of serum vibriocidal antibody (SVA) against the classical Inaba biotype of V. cholerae at Day 11 following one dose of VAXCHORA, defined as a 4-fold or greater rise over baseline Day 1 SVA titer
Time Frame: Day 11
Population: Immunogenicity Evaluable Population (IEP)
Measure: Number (98.3% Confidence Interval); unit: percentage of participants
Groups:
- Cohort 1 (Placebo, 12-17 Yrs): Subjects aged 12 - 17 were administered a 100 mL oral dose of placebo on Day 1, and had study visits on Day 11, 29, 91 and 181.
Arm/Group | Cohort 1 (Active, 12-17 Yrs) | Cohort 1 (Placebo, 12-17 Yrs)
Number analyzed (Participants) | 157 | 23
percentage of participants | 99.4 [95.4 to 99.9] | 0 [0.0 to 14.3]
Statistical Analysis 1: Comparison: Cohort 1 (Active, 12-17 Yrs); Test type: Non-Inferiority — This analysis was based on the lower confidence limit and did not entail a comparative group. The requirement was for the lower limit of the 98.3% CI be at least 70%. Multiplicity adjustment due to co-primary endpoints allotted alpha=0.017 to this endpoint resulting in a 98.3% confidence interval; Proportion = 0.985, 98.3% CI 1-sided [lower limit 0.7]

2. Primary Outcome: Cohort 2 (6 to <12 Years) Primary Endpoint - Seroconversion of Serum Vibriocidal Antibody Against V. Cholerae
Description: as for outcome 1
Time Frame: Day 11
Population: Immunogenicity Evaluable Population (IEP)
Measure: Number (98.3% Confidence Interval); unit: percentage of participants
Groups:
- Cohort 2 (Placebo, 6-11 Yrs): Subjects aged 6 - 11 were administered a 100 mL oral dose of placebo on Day 1, and had study visits on Day 11, 29, 91 and 181.
Arm/Group | Cohort 2 (Active, 6 - 11 Yrs) | Cohort 2 (Placebo, 6-11 Yrs)
Number analyzed (Participants) | 139 | 24
percentage of participants | 97.8 [92.5 to 99.4] | 4.2 [0.7 to 20.2]
Statistical Analysis 1: Comparison: Cohort 2 (Active, 6 - 11 Yrs) vs Cohort 2 (Placebo, 6-11 Yrs); Test type: Non-Inferiority — This analysis was based on the lower confidence limit and did not entail a comparative group. The requirement was for the lower limit of the 98.3% CI be at least 70%. Multiplicity adjustment due to coprimary endpoints allotted alpha=0.017 to this endpoint resulting in a 98.3% confidence interval; Proportion = 0.985, 98.3% CI 1-sided [lower limit 0.7]

3. Primary Outcome: Cohort 3 (2 to <6 Years) Primary Endpoint - Seroconversion of Serum Vibriocidal Antibody Against V. Cholerae
Description: as for outcome 1
Time Frame: Day 11
Population: Immunogenicity Evaluable Population (IEP)
Measure: Number (98.3% Confidence Interval); unit: percentage of participants
Groups:
- Cohort 3 (Placebo, 2-5 Yrs): Subjects aged 2 - 5 were administered a 50 mL oral dose of placebo on Day 1, and had study visits on Day 11, 29, 91 and 181.
Arm/Group | Cohort 3 (Active, 2 - 5 Yrs) | Cohort 3 (Placebo, 2-5 Yrs)
Number analyzed (Participants) | 103 | 20
percentage of participants | 98.1 [91.5 to 99.6] | 0 [0.0 to 16.1]
Statistical Analysis 1: Comparison: Cohort 3 (Active, 2 - 5 Yrs) vs Cohort 3 (Placebo, 2-5 Yrs); Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Proportion = 0.985, 98.3% CI 1-sided [lower limit 0.7]

4. Primary Outcome: Cohort 1 (12-17 Yrs) Primary Endpoint - Non-inferiority of Seroconversion Rate at Day 11 Relative to Adults Aged 18 - 45 Years
Description: The seroconversion rate is defined as the percentage of subjects with a 4-fold or greater rise over baseline Day 1 Serum Vibriocidal Antibody (SVA) titer against the classical Inaba biotype of V. cholerae at Day 11 following one dose of Vaxchora vaccine. The hypothesis was that the pediatric seroconversion rate would be non-inferior to the seroconversion rate at Day 11 in adults between the ages of 18 and 45 years.
Time Frame: Day 11
Population: Immunogenicity Evaluable Population (IEP)
Measure: Number (98.3% Confidence Interval); unit: percentage of participants
Groups:
- Historical Control: Adult Bridging Population: This arm consists of historical data from Vaxchora vaccine subjects from study PXVX-VC-200-004. The data was included in study PXVX-VC-200-006 as a comparator bridging population for the Day 11 seroconversion.
Arm/Group | Cohort 1 (Active, 12-17 Yrs) | Historical Control: Adult Bridging Population
Number analyzed (Participants) | 157 | 2687
percentage of participants | 99.4 [95.4 to 99.9] | 93.5 [92.3 to 94.6]
Statistical Analysis 1: Comparison: Cohort 1 (Active, 12-17 Yrs) vs Historical Control: Adult Bridging Population; Test type: Non-Inferiority — Non-inferiority was determined using the Newcombe method of determining the difference between two independent binomial distributions. Multiple comparison adjustment for co-primary endpoints allotted alpha=0.033 to this comparison. The lower limit of the 96.7% CI needed to be greater than -10 percentage points to prove non-inferiority; Risk Difference (RD) = 5.8, 96.7% CI 2-sided [2.4 to 7.1] — Newcombe method of determining the difference between two independent binomial distributions

5. Primary Outcome: Cohort 2 (6-11 Yrs) Primary Endpoint - Non-inferiority of Seroconversion Rate at Day 11 Relative to Adults Aged 18 - 45 Years
Description: as for outcome 4
Time Frame: Day 11
Population: Immunogenicity Evaluable Population (IEP)
Measure: Number (98.3% Confidence Interval); unit: percentage of participants
Groups:
- Cohort 2 (Active, 6-11 Yrs): Subjects aged 6 - 11 were administered a 100 mL oral dose of Vaxchora vaccine on Day 1, and had study visits on Day 11, 29, 91 and 181.
  VAXCHORA (Cholera Vaccine, Live, Oral): VAXCHORA (Cholera Vaccine, Live, Oral) is a live, attenuated bacterial vaccine suspension for oral administration containing the V. cholerae strain CVD 103-HgR.
Arm/Group | Cohort 2 (Active, 6-11 Yrs) | Historical Control: Adult Bridging Population
Number analyzed (Participants) | 139 | 2687
percentage of participants | 97.8 [92.5 to 99.4] | 93.5 [92.3 to 94.6]
Statistical Analysis 1: Comparison: Cohort 2 (Active, 6-11 Yrs) vs Historical Control: Adult Bridging Population; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; Risk Difference (RD) = 4.3, 96.7% CI 2-sided [-0.3 to 6.2]

6. Primary Outcome: Cohort 3 (2-5 Yrs) Primary Endpoint - Non-inferiority of Seroconversion Rate at Day 11 Relative to Adults Aged 18 - 45 Years
Description: The seroconversion rate is defined as the percentage of subjects with a 4-fold or greater rise over baseline Day 1 Serum Vibriocidal Antibody (SVA) titer against the classical Inaba biotype of V. cholerae at Day 11 following one dose of Vaxchora vaccine. The hypothesis was that the pediatric seroconversion rate would be non-inferior to the seroconversion rate at Day 11 in adults between the ages of18 and 45 years.
Time Frame: Day 11
Population: Immunogenicity Evaluable Population (IEP)
Measure: Number (98.3% Confidence Interval); unit: percentage of participants
Groups:
- Cohort 3 (Active, 2-5 Yrs): Subjects aged 2 - 5 were administered a 50 mL oral dose of Vaxchora vaccine on Day 1, and had study visits on Day 11, 29, 91 and 181.
  VAXCHORA (Cholera Vaccine, Live, Oral): VAXCHORA (Cholera Vaccine, Live, Oral) is a live, attenuated bacterial vaccine suspension for oral administration containing the V. cholerae strain CVD 103-HgR.
Arm/Group | Cohort 3 (Active, 2-5 Yrs) | Historical Control: Adult Bridging Population
Number analyzed (Participants) | 103 | 2687
percentage of participants | 98.1 [91.5 to 99.6] | 93.5 [92.3 to 94.6]
Statistical Analysis 1: Comparison: Cohort 3 (Active, 2-5 Yrs) vs Historical Control: Adult Bridging Population; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; Risk Difference (RD) = 4.5, 96.7% CI 2-sided [-1.1 to 6.4]

7. Secondary Outcome: Cohort 1 (12 to <18 Years) - Seroconversion of SVA - Day 29
Description: Seroconversion of SVA against the classical Inaba biotype of V. cholerae at Day 29 for all subjects
Time Frame: Day 29
Population: Immunogenicity Evaluable Population (IEP)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 (Active, 12-17 Yrs) | Cohort 1 (Placebo, 12-17 Yrs)
Number analyzed (Participants) | 156 | 23
percentage of participants | 100 [97.6 to 100] | 0 [0.0 to 14.3]
Statistical Analysis 1: Comparison: Cohort 1 (Active, 12-17 Yrs) vs Cohort 1 (Placebo, 12-17 Yrs); Test type: Superiority — Fisher's exact test was used to compare Vaxchora vaccine to placebo on the percent of subjects who seroconverted. For Vaxchora vs placebo within each cohort at each Day on study timepoint, the p-value was the same (p<0.0001); p < 0.0001, Fisher Exact

8. Secondary Outcome: Cohort 1 (12 to <18 Years) - Seroconversion of SVA - Day 91
Description: Seroconversion of SVA against the classical Inaba biotype of V. cholerae at Day 91 for all subjects
Time Frame: Day 91
Population: Immunogenicity Evaluable Population (IEP)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 (Active, 12-17 Yrs) | Cohort 1 (Placebo, 12-17 Yrs)
Number analyzed (Participants) | 156 | 23
percentage of participants | 85.6 [79.2 to 90.3] | 0 [0.0 to 14.3]
Statistical Analysis 1: Comparison: Cohort 1 (Active, 12-17 Yrs) vs Cohort 1 (Placebo, 12-17 Yrs); Test type: Superiority — [test comment as in outcome 7, analysis 1]; p < 0.0001, Fisher Exact

9. Secondary Outcome: Cohort 1 (12 to <18 Years) - Seroconversion of SVA - Day 181
Description: Seroconversion of SVA against the classical Inaba biotype of V. cholerae at Day 181 for all subjects
Time Frame: Day 181
Population: Immunogenicity Evaluable Population (IEP)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 (Active, 12-17 Yrs) | Cohort 1 (Placebo, 12-17 Yrs)
Number analyzed (Participants) | 156 | 23
percentage of participants | 73.5 [66.0 to 79.9] | 0 [0.0 to 15.5]
Statistical Analysis 1: Comparison: Cohort 1 (Active, 12-17 Yrs) vs Cohort 1 (Placebo, 12-17 Yrs); Test type: Superiority — [test comment as in outcome 7, analysis 1]; p < 0.0001, Fisher Exact

10. Secondary Outcome: Cohort 1 (12 to <18 Years) - Seroconversion of SVA - Day 365
Description: Seroconversion of SVA against the classical Inaba biotype of V. cholerae at Day 365 for all subjects
Time Frame: Day 365
Population: Immunogenicity Evaluable Population (IEP)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 (Active, 12-17 Yrs)
Number analyzed (Participants) | 70
percentage of participants | 68.6 [57.0 to 78.2]

11. Secondary Outcome: Cohort 1 (12 to <18 Years) - Seroconversion of SVA - Day 547
Description: Seroconversion of SVA against the classical Inaba biotype of V. cholerae at Day 547 for all subjects
Time Frame: Day 547
Population: Immunogenicity Evaluable Population (IEP)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 (Active, 12-17 Yrs)
Number analyzed (Participants) | 67
percentage of participants | 73.1 [61.5 to 82.3]

12. Secondary Outcome: Cohort 1 (12 to <18 Years) - Seroconversion of SVA - Day 730
Description: Seroconversion of SVA against the classical Inaba biotype of V. cholerae at Day 730 for all subjects
Time Frame: Day 730
Population: Immunogenicity Evaluable Population (IEP)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 (Active, 12-17 Yrs)
Number analyzed (Participants) | 62
percentage of participants | 64.5 [52.1 to 75.3]

13. Secondary Outcome: Cohort 2 (6 to <12 Years) - Seroconversion of SVA - Day 29
Description: Seroconversion of SVA against the classical Inaba biotype of V. cholerae at Day 29 for all subjects
Time Frame: Day 29
Population: Immunogenicity Evaluable Population (IEP)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2 (Active, 6 - 11 Yrs) | Cohort 2 (Placebo, 6-11 Yrs)
Number analyzed (Participants) | 138 | 23
percentage of participants | 94.9 [89.9 to 97.5] | 4.3 [0.8 to 21.0]
Statistical Analysis 1: Comparison: Cohort 2 (Active, 6 - 11 Yrs) vs Cohort 2 (Placebo, 6-11 Yrs); Test type: Superiority — [test comment as in outcome 7, analysis 1]; p < 0.0001, Fisher Exact

14. Secondary Outcome: Cohort 3 (2 to <6 Years) - Seroconversion of SVA - Day 29
Description: Seroconversion of SVA against the classical Inaba biotype of V. cholerae at Day 29 for all subjects
Time Frame: Day 29
Population: Immunogenicity Evaluable Population (IEP)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 3 (Active, 2 - 5 Yrs) | Cohort 3 (Placebo, 2-5 Yrs)
Number analyzed (Participants) | 98 | 18
percentage of participants | 93.9 [87.3 to 97.2] | 0 [0.0 to 17.6]
Statistical Analysis 1: Comparison: Cohort 3 (Active, 2 - 5 Yrs) vs Cohort 3 (Placebo, 2-5 Yrs); Test type: Superiority — [test comment as in outcome 7, analysis 1]; p < 0.0001, Fisher Exact

15. Other Pre Specified Outcome: Cohort 1 (12 to <18 Years) Exploratory Endpoint - Anti-O1 Lipopolysaccharide Memory B Cell Concentration at Day 1
Description: Anti-O1 lipopolysaccharide (LPS) memory B cell concentration at Day 1 for the subjects in the active treatment group and the placebo crossover group
Time Frame: Day 1
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Cohort 1 (12 to <18 Years) Exploratory Endpoint - Anti-O1 Lipopolysaccharide Memory B Cell Concentration at Day 91
Description: Anti-O1 lipopolysaccharide (LPS) memory B cell concentration at Day 91 for the subjects in the active treatment group and the placebo crossover group
Time Frame: Day 91
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Cohort 1 (12 to <18 Years) Exploratory Endpoint - Anti-O1 Lipopolysaccharide Memory B Cell Concentration at Day 181
Description: Anti-O1 lipopolysaccharide (LPS) memory B cell concentration at Day 181 for the subjects in the active treatment group and the placebo crossover group
Time Frame: Day 181
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Cohort 1 (12 to <18 Years) Exploratory Endpoint - Anti-O1 Lipopolysaccharide Memory B Cell Concentration at Day 365
Description: Anti-O1 lipopolysaccharide (LPS) memory B cell concentration at Day 365 for the subjects in the active treatment group who participate in the substudy.
Time Frame: Day 365
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Cohort 1 (12 to <18 Years) Exploratory Endpoint - Anti-O1 Lipopolysaccharide Memory B Cell Concentration at Day 547
Description: Anti-O1 lipopolysaccharide (LPS) memory B cell concentration at Day 547 for the subjects in the active treatment group who participate in the substudy.
Time Frame: Day 547
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Cohort 1 (12 to <18 Years) Exploratory Endpoint - Anti-O1 Lipopolysaccharide Memory B Cell Concentration at Day 730
Description: Anti-O1 lipopolysaccharide (LPS) memory B cell concentration at Day 730 for the subjects in the active treatment group who participate in the substudy.
Time Frame: Day 730
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Safety - Solicited Adverse Events
Description: Evaluate the safety and tolerability of VAXCHORA by collecting solicited adverse events (abdominal pain, headache, lack of appetite, tiredness, diarrhea, nausea, vomiting and fever) by age cohort and overall through Day 8
Time Frame: Through Day 8
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Safety - Unsolicited Adverse Events
Description: Evaluate the safety and tolerability of VAXCHORA by collecting unsolicited adverse events by age cohort and overall through Day 29
Time Frame: Through Day 29
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Safety - Serious Adverse Events
Description: Evaluate the safety and tolerability of VAXCHORA by collecting serious adverse events by age cohort and overall through Day 181
Time Frame: Through Day 181
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Acceptability
Description: Evaluate the acceptability of VAXCHORA using the percent of subjects in each age cohort able to complete the dosing according to protocol.
Time Frame: Day 1
Population: The data presented is for the population that was randomized and received treatment. For Cohort 2, 2 Vaxchora subjects and 1 placebo subject were randomized, but not treated. For Cohort 3, 4 Vaxchora subjects were randomized, but not treated.
Measure: Number; unit: percent of participants
Arm/Group | Cohort 1 (Active, 12-17 Yrs) | Cohort 1 (Placebo, 12 - 17 Yrs) | Cohort 2 (Active, 6 - 11 Yrs) | Cohort 2 (Placebo, 6 - 11 Yrs) | Cohort 3 (Active, 2 - 5 Yrs) | Cohort 3 (Placebo, 2 - 5 Yrs)
Number analyzed (Participants) | 163 | 26 | 156 | 26 | 146 | 26
percent of participants | 99.4 | 100 | 91.0 | 96.2 | 79.5 | 73.1

ADVERSE EVENTS:
Time Frame: All adverse events were collected for 28 days post vaccination. Serious adverse events were followed until the end of the end of the subject's participation in the study (2 years for adolescents in the long term sub-study and 6 months for all others). Solicited adverse events were collected for daily for 8 consecutive days following vaccination (Days 1-8). Events that continued past Day 8 were recorded as unsolicited adverse events.
Description: The Historical Control population is not included in this section as comparisons between the pediatric and adult populations were not specified to be conducted in the protocol.
  The data below is not for randomized subjects, but for those included in the safety population.
  For cohort 1, 2 subjects received Vaxchora instead of placebo; the subject count is 165 Vaxchora : 24 placebo.
  For cohort 2, 1 subject received Vaxchora instead of placebo; the subject count is 157 Vaxchora : 25 placebo.
Arm/Group | Cohort 1 (Active, 12-17 Yrs) | Cohort 1 (Placebo, 12 - 17 Yrs) | Cohort 2 (Active, 6 - 11 Yrs) | Cohort 2 (Placebo, 6 - 11 Yrs) | Cohort 3 (Active, 2 - 5 Yrs) | Cohort 3 (Placebo, 2 - 5 Yrs)
All-Cause Mortality (participants affected / at risk) | 0/165 | 0/24 | 0/157 | 0/25 | 0/146 | 0/26
Serious Adverse Events (participants affected / at risk) | 4/165 | 0/24 | 0/157 | 0/25 | 0/146 | 1/26
Other Adverse Events (participants affected / at risk) | 116/165 | 13/24 | 93/157 | 15/25 | 74/146 | 12/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (Active, 12-17 Yrs) (N=165) | Cohort 1 (Placebo, 12 - 17 Yrs) (N=24) | Cohort 2 (Active, 6 - 11 Yrs) (N=157) | Cohort 2 (Placebo, 6 - 11 Yrs) (N=25) | Cohort 3 (Active, 2 - 5 Yrs) (N=146) | Cohort 3 (Placebo, 2 - 5 Yrs) (N=26)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intentional Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Local Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (Active, 12-17 Yrs) (N=165) | Cohort 1 (Placebo, 12 - 17 Yrs) (N=24) | Cohort 2 (Active, 6 - 11 Yrs) (N=157) | Cohort 2 (Placebo, 6 - 11 Yrs) (N=25) | Cohort 3 (Active, 2 - 5 Yrs) (N=146) | Cohort 3 (Placebo, 2 - 5 Yrs) (N=26)
Abdominal Pain (Gastrointestinal disorders) | 62 (130) | 4 (10) | 43 (83) | 6 (15) | 25 (53) | 4 (7) — Solicited Day 1 - 8
Headache (Nervous system disorders) | 74 (191) | 11 (18) | 41 (77) | 6 (11) | 13 (18) | 2 (3) — Solicited Day 1 - 8
Lack of Appetite (Metabolism and nutrition disorders) | 48 (112) | 3 (8) | 24 (47) | 5 (11) | 28 (63) | 3 (8) — Solicited Day 1 - 8
Fatigue (General disorders) | 67 (170) | 9 (30) | 55 (123) | 8 (17) | 45 (108) | 6 (13) — Solicited Day 1 - 8
Diarrhea (Gastrointestinal disorders) | 6 (7) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Solicited Day 1 - 8
Nausea (Gastrointestinal disorders) | 37 (69) | 6 (16) | 22 (37) | 4 (11) | 10 (14) | 4 (4) — Solicited Day 1 - 8
Vomiting (Gastrointestinal disorders) | 9 (14) | 0 (0) | 7 (12) | 0 (0) | 2 (2) | 3 (3) — Solicited Day 1 - 8
Fever (General disorders) | 3 (4) | 0 (0) | 5 (6) | 1 (1) | 3 (4) | 1 (3) — Solicited Day 1 - 8
Headache (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unsolicited Day 29
Lack of Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) — Unsolicited Day 29
Fatigue (General disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) — Unsolicited Day 29
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Unsolicited Day 29
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) — Unsolicited Day 29
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unsolicited Day 29
Joint Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unsolicited Day 29
Arthropod Bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Unsolicited Day 29
Vessel Puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unsolicited Day 29
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unsolicited Day 29
Loose Stool (Gastrointestinal disorders) | 23 (30) | 5 (6) | 18 (19) | 0 (0) | 8 (8) | 2 (2) — Unsolicited Day 29
Rectal Tenesmus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unsolicited Day 29
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unsolicited Day 29
Upper Respiratory Tract Infection (Infections and infestations) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 3 (3) — Unsolicited Day 29
Furuncle (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unsolicited Day 29
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) — Unsolicited Day 29
Otitis Media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unsolicited Day 29
Ear Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) — Unsolicited Day 29
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Unsolicited Day 29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/37/NCT03220737/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/37/NCT03220737/SAP_001.pdf